CLINICAL TRIAL: NCT05902351
Title: Global Registry for Inherited Neuropathies Natural History Study for Charcot Marie Tooth Disease
Brief Title: Natural History Study for Charcot Marie Tooth Disease
Status: Recruiting | Type: Observational
Sponsor: Hereditary Neuropathy Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: GRIN1001
Record Dates: First submitted 2023-05-02; First posted 2023-06-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Charcot-Marie-Tooth Disease; Charcot-Marie-Tooth; Charcot-Marie-Tooth Disease, Type IA; Charcot-Marie-Tooth Disease Type 2A; Charcot-Marie-Tooth Disease Type 2; Charcot-Marie-Tooth Disease, Type 2C; Charcot-Marie-Tooth Disease Type 2A2B; Charcot-Marie-Tooth Disease Type 2B2; Charcot-Marie-Tooth Disease Type 2A1; Charcot-Marie-Tooth Disease Type 4B1; Charcot-Marie-Tooth Disease, Type IB; Charcot-Marie-Tooth Disease Type 2B1; Charcot-Marie-Tooth Disease Type 2U (Diagnosis); Charcot-Marie-Tooth Disease Type 4A; Charcot-Marie-Tooth Disease, Type 4A, Axonal Form; Charcot-Marie-Tooth Disease Type 2A2A; Charcot-Marie-Tooth Disease Type 2S (Disorder); Charcot-Marie-Tooth Disease and Deafness; Charcot-Marie-Tooth Disease Type 4B2; Charcot-Marie-Tooth Disease Type 4H; Charcot-Marie-Tooth Disease Type 1F; Charcot-Marie-Tooth Disease Type 4C; Charcot-Marie-Tooth Disease Type 4E; Charcot-Marie-Tooth Disease Type 1D; Charcot-Marie-Tooth Disease Type 2Q (Diagnosis); Charcot-Marie-Tooth Disease Type 2A2; Charcot-Marie-Tooth Disease Type 2N (Diagnosis); Charcot-Marie-Tooth Disease Type 2B5; Charcot-Marie-Tooth Disease Type 2D; Charcot-Marie-Tooth Disease Type 4D; Charcot-Marie-Tooth Disease Type 2K; Charcot-Marie-Tooth Disease Type 2L (Diagnosis); Charcot-Marie-Tooth Disease Type 2T; Charcot-Marie-Tooth Disease Type 2I; Charcot-Marie-Tooth Disease Type 2J; Charcot-Marie-Tooth Disease Type 2E; Charcot-Marie-Tooth Disease Type 2G; Charcot-Marie-Tooth Disease Type 1C; Charcot-Marie-Tooth Disease Type 2R; Charcot-Marie-Tooth Disease Type 2O (Diagnosis); Charcot-Marie-Tooth Disease Type 2M; Charcot-Marie-Tooth Disease Type 2P; Charcot-Marie-Tooth Disease Type 2Y; Charcot-Marie-Tooth Disease Type 4F (Diagnosis); Charcot-Marie-Tooth Disease Type 4B3; Charcot-Marie-Tooth Disease Type 2H; HNPP; X-Linked Charcot-Marie-Tooth Disease
Keywords: Inherited Neuropathies; Peripheral Neuropathy; Charcot-Marie-Tooth; Charcot-Marie-Tooth Disease; CMT
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Charcot-Marie-Tooth disease, Type 2A; Charcot-Marie-Tooth disease, Type 2C; Charcot-Marie-Tooth disease, Type 2B2; Charcot-Marie-Tooth Disease, Axonal, Type 2a1; Charcot-Marie-Tooth disease, Type 4B1; Limb-girdle muscular dystrophy, type 1B; Disease; Charcot-Marie-Tooth disease, Type 4A; Charcot-Marie-Tooth disease, Type 4A, axonal form; Charcot-Marie-Tooth Disease, Axonal, Type 2A2; Charcot-Marie-Tooth disease and deafness; Charcot-Marie-Tooth disease, Type 4B2; Charcot-Marie-Tooth Disease, Type 4H; Charcot-Marie-Tooth disease, Type 1F; Charcot-Marie-Tooth disease, Type 4C; Charcot-Marie-Tooth disease, Type 4E; Charcot-Marie-Tooth disease, Type 1D; Charcot-Marie-Tooth Disease, Axonal, Type 2n; Charcot-Marie-Tooth disease, Type 2D; Neuropathy, hereditary motor and sensory, LOM type; Charcot-Marie-Tooth disease, Type 2K; Charcot-Marie-Tooth disease, Type 2I; Charcot-Marie-Tooth disease, Type 2J; Charcot-Marie-Tooth disease, Type 2E; Charcot-Marie-Tooth disease, Type 2H; Charcot-Marie-Tooth disease, Type 1C; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this Natural History Study for Charcot-Marie-Tooth is to acquire, record, and analyze patient-reported data and associated genetic reports, Electronic Health Records (EHRs) and clinical notes to identify the burden, diagnostic journey, and prevalence of disease that will aid scientists in their work toward finding a cure.

Participants will be asked to complete a Natural History Survey.

ELIGIBILITY:
Inclusion Criteria:

Patients will be made aware of the study by HNF and others (referenced above) and invited to participate. Once patients have reviewed and signed electronically the informed consent document, it is attached to their file.

All affected individuals with CMT/IN are eligible to participate in GRIN with proper informed consent.

Children, adolescents and adults with either a confirmed diagnosis or suspected to have CMT/IN are eligible with parent and/or guardian consent.

Individuals that have been clinically diagnosed through family history and/or standard clinical testing (e.g. neuro exam, EMG, NCS) and/or genetically tested or suspected to have CMT/IN (note: many mutations have not been identified yet) are eligible.

Exclusion Criteria:

People that do not have Charcot-Marie-Tooth or other Inherited Neuropathies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is open to anyone that has Charcot-Marie-Tooth Disease or other Inherited Neuropathies.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify the type of CMT | 156 weeks
  Patient-Reported Outcomes depending on individual experience I.e. Genetic testing, clinical observation, EMG, family history.
Disease Symptoms | 156 weeks
  Patient-Reported Observations
Impact of symptoms on Activities of Daily Living | 156 weeks
  Patient-Reported Observations
Associated Comorbidities | 156 weeks
  Patient-Reported Observations

CONTACTS AND LOCATIONS:
Overall Officials: Allison Moore, Principal Investigator — Hereditary Neuropathy Foundation
Locations (1):
- Hereditary Neuropathy Foundation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Landing page and entry for patients to participate in the Global Registry for Inherited Neuropathies — https://www.hnf-cure.org/cmt/cmt-research/grin-patient-registry/